CLINICAL TRIAL: NCT04937101
Title: Human Subject Research Ethics Committee, 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Brief Title: The Safety and Effectiveness of Local Injection of Antihistamines in Treatment of Inflammatory Skin Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-837
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-01

CONDITIONS: Inflammatory Skin Disease
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antihistamine treatment group (Experimental): Chlorpheniramine, the concentration is 10mg/ml per unit point, the highest dose is 1ml
  Interventions: Drug: Chlorpheniramine-Codeine
- Control group (No Intervention)

INTERVENTIONS:
Drug: Chlorpheniramine-Codeine — When the filter tester is sensitive, he opened the random letter group envelope to the notification letter manager and jointly confirmed the classification of the message group. The test group used the chlorpheniramine beacon, the physiological surface was used, and the local lesions of fine particles were used in the focus. Injection therapy. No form of anesthesia is used during injection. A total of injection treatment, at intervals, each treatment and the last treatment, treatment and safety after 1 month.
  Arms: Antihistamine treatment group

SUMMARY:
The treatment of chronic inflammatory skin diseases is a difficult point in clinical diseases, which mainly include patients with pathological scars, sarcoidosis and chronic eczema. Chronic nodular lesions and long-term itching symptoms bring great physical and mental pain to patients.

Long-term repeated treatments are required. At present, the most commonly used treatment is intralesional injection of glucocorticoids. Long-term glucocorticoid injections have some side effects, including pain, hypopigmentation, skin atrophy, pigmentation, telangiectasia and menstrual disorders in women. There are a large number of clinical patients who still lack safe and effective drugs, including children, pregnant women, patients with weakened or defective immunity, and even patients with mild inflammatory skin diseases with mainly itching symptoms.

The systemic and topical application of antihistamine drugs provides new ideas for the treatment of inflammatory skin. As the most commonly used clinical antihistamine, chlorpheniramine has a long history in the treatment of allergic diseases and can improve the body's inflammatory state. At the same time, the drug has high safety and is suitable for children and pregnant women, or patients with underlying diseases such as hypertension, diabetes, and immunodeficiency diseases.

DETAILED DESCRIPTION:
At present, there are more and more reports about the application of antihistamines to the treatment of pathological scars. Exposing fibroblasts from normal skin and keloids to the antihistamine diphenhydramine can inhibit the growth of keloid fibroblasts . Based on the existing research foundation in the field and the results of our previous laboratory experiments, we hypothesize that intralesional injection of chlorpheniramine can improve the pruritus symptoms and the severity of skin lesions in inflammatory skin diseases, and can be used as a new application of traditional medicine.

ELIGIBILITY:
Inclusion criteria 1. Meet the diagnostic criteria of chronic inflammatory skin disease, with limited lesions, mainly including pathological scars, isolated lesions of sarcoidosis and local hypertrophic lesions of chronic eczema; 2. Good compliance, agree not to accept the test during the test period Any local injection treatment other than treatment; 3. Voluntarily sign an informed consent form and agree to participate in all visits, inspections and treatments in accordance with the requirements of the trial protocol.

Exclusion criteria

1. Those who have received triamcinolone acetonide injection treatment in the lesion area within the past year; 2. Those who have precancerous skin lesions or have a tendency to become cancerous, or those who have received local radiation therapy on their skin; 3. There are skin infections, inflammations, herpes, and silver Those with active skin diseases such as scaly; 4. Those who have autoimmune diseases or are receiving immunotherapy; 5. Those who have coagulation dysfunction or are using anticoagulant/antiplatelet drugs; 6. Those who have other serious diseases, such as liver and kidney Insufficiency, diabetes, high blood pressure, etc.; 7. Women who are planning to become pregnant, pregnant or breastfeeding; 8. People who suffer from mental illness, or are currently taking antipsychotic drugs; 9. Other conditions that the investigator considers inappropriate to participate in this trial , Such as high expectations, poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The degree of improvement in lesion thickness | 1 year
  After a treatment cycle of the lesion, the degree of improvement in the thickness of the lesion is graded according to the total score of the patient's self-evaluation and the doctor's evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Huan Qian, MD, Principal Investigator — 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided